CLINICAL TRIAL: NCT02201017
Title: HeartTrends HRV Algorithm for the Detection of Myocardial Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-1194-IG-CTIL
Record Dates: First submitted 2014-07-16; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Heart Rate Variability Ischemia Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A total of 621 consecutive male and female subjects, without established CAD, referred to exercise stress testing (EST) due to 1) chest pain syndromes or equivocal/equivalent angina with intermediate pretest probability for CAD; 2) , or asymptomatic subjects with diabetes mellitus who are referred EST for risk assessment prior to initiation of an exercise program.

To validate the diagnostic performance of the HeartTrends device for the detection and ruling out of myocardial ischemia in a population of subjects who are currently referred for cardiovascular evaluation using EST.

Prospective multicenter single-armed study, assessing the diagnostic accuracy of HRV analysis by the HeartTrends device for the detection of myocardial ischemia, as determined by stress echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* No known CAD
* Referral for EST due to either one of the following two indications:

  1. Chest pain syndrome or equivocal angina in subjects with intermediate pretest probability of CAD according to the 2002 updated guidelines for exercise stress examination.1 (See definition of intermediate pretest probability of CAD in Supplementary Appendix Table at the end of this document); or
  2. Asymptomatic subjects with diabetes mellitus referred to EST for risk assessment prior to initiation of an exercise program.
* Willing and able to provide written informed consent

Exclusion Criteria:

1. Acute Coronary Syndrome
2. Established CAD
3. Atrial fibrillation or flutter
4. Cardiac Pacemaker
5. Clinical diagnosis of heart failure
6. Severe COPD (FEV1< 50% predicted value)
7. Active myocarditis, constrictive pericarditis, any cardiomyopathy, cardiac or systemic amyloidosis
8. Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
9. Any illness that might reduce life expectancy to less than 1 year from screening
10. Left bundle branch block (LBBB), significant intra-ventricular conduction delay (IVCD) or significant (>1mm) ST deviations on baseline ECG
11. Inability to perform an exercise stress test (i.e. orthopedical or neurological limitations)
12. Any significant valvular disease defined as:

Established valvular regurgitation or stenosis abnormality above moderate severity 13. BMI >35 kg/m2 14. Recent (< 6 months) history of pulmonary embolism

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 621 consecutive male and female subjects, without established CAD, referred to exercise stress testing (EST) due to 1) chest pain syndromes or equivocal/equivalent angina with intermediate pretest probability for CAD; 2) , or asymptomatic subjects with diabetes mellitus who are referred EST for risk assessment prior to initiation of an exercise program.
  Pretest probability of CAD will be based on the ACC 2002 guideline update on exercise stress testing1.
Sampling Method: Non-Probability Sample
Enrollment: 621 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Positive percent agreement | 1 year
  Positive percent agreement of ≥70% (with a lower confidence interval of 60%) between a positive HRV HeartTrends test and a positive ESE

SECONDARY OUTCOMES:
negative percent agreement | 1 year
  HeartTrends device testing is associated with a negative percent agreement of ≥70% with negative results detected by ESE.
  ≥10% difference between the positive percent agreement of HRV with ESE and the positive percent agreement of EST with ESE.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, MD, Study Director — THE ISRAELI ASSOCIATION FOR CARDIOVASCULAR TRIALS
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Sheba medical center, Ramat Gan, Israel

REFERENCES:
- [Derived] Goldenberg I, Goldkorn R, Shlomo N, Einhorn M, Levitan J, Kuperstein R, Klempfner R, Johnson B. Heart Rate Variability for Risk Assessment of Myocardial Ischemia in Patients Without Known Coronary Artery Disease: The HRV-DETECT (Heart Rate Variability for the Detection of Myocardial Ischemia) Study. J Am Heart Assoc. 2019 Dec 17;8(24):e014540. doi: 10.1161/JAHA.119.014540. Epub 2019 Dec 16. PMID 31838969